CLINICAL TRIAL: NCT01830101
Title: A Randomized Phase III Study of Re-Irradiation in Recurrent Glioblastoma
Brief Title: A Phase III Study of Re-Irradiation in Recurrent Glioblastoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This study will not be proceeding due to lack of funding from anticipated sources
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCI-Patel-01
Record Dates: First submitted 2013-03-13; First posted 2013-04-12 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2014-02

CONDITIONS: Recurrent Glioblastoma
Keywords: recurrent glioblastoma; re-irradiation; continuous low-dose temozolomide
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TMZ plus concurrent re-irradiation (Experimental): TMZ plus concurrent re-irradiation
  Interventions: Drug: TMZ plus concurrent re-irradiation; Drug: Temozolomide
- TMZ alone (Experimental): TMZ alone
  Interventions: Drug: TMZ plus concurrent re-irradiation; Drug: Temozolomide

INTERVENTIONS:
Drug: TMZ plus concurrent re-irradiation
  Other Names: Temedol
Drug: Temozolomide — low-dose temozolomide daily for one year
  Other Names: Temedol

SUMMARY:
The investigators hope to improve overall median survival of patients with recurrent Glioblastoma by investigating continuous low-dose daily Temozolomide plus or minus five treatments of re-irradiation.

DETAILED DESCRIPTION:
This is a stratified study for patients with recurrent intracranial glioblastoma or gliosarcoma previously treated with concurrent chemoradiation presenting radiographic progression or recurrence of tumour. Patients are stratified by extent of resection, time to re-irradiation and re-irradiation volume.

ELIGIBILITY:
Inclusion Criteria:

* histologically-proven intracranial glioblastoma or gliosarcoma previously treated with concurrent chemoradiation
* radiographic evidence of tumour progression or recurrence
* 18 years or older
* ECOG 0 - 2
* signed informed consent form

Exclusion Criteria:

* tumour progression or recurrence within 3 months of initial concurrent chemoradiation
* 6 or more cycles of TMZ administered following chemoradiation at initial diagnosis
* more than one prior course of salvage chemo for recurrent disease
* prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for greater or equal to 3 years
* prior head or neck RT except for T1 glottic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
To determine the overall median survival of the combination of continuous dose-intense temozolomide with or without re-irradiation in patients with recurrent glioblastoma. | 2 months

SECONDARY OUTCOMES:
To evaluate time to radiographic progression or recurrence of tumour following treatment with continuous dose-intense temozolomide with or without re-irradiation. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Samir Patel, MD, Principal Investigator — Cross Cancer Institute; Gerald Lim, MD, Principal Investigator — Tom Baker Cancer Centre
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada